CLINICAL TRIAL: NCT01773512
Title: The Prediction of Extent and Risk Profile of Coronary Atherosclerosis (Examined by Intravascular Ultrasound, Virtual Histology and Optical Coherence Tomography) and Their Changes During Lipid-lowering Therapy Based on Non-invasive Techniques.
Brief Title: The Prediction of Extent and Risk Profile of Coronary Atherosclerosis and Their Changes During Lipid-lowering Therapy Based on Non-invasive Techniques
Acronym: PREDICT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: General University Hospital, Prague (Other)
Collaborators: Ministry of Health, Czech Republic (Other Government); Czech Ministry of Education (Other Government); University of Iowa (Other); Loyola University Chicago (Other)
Responsible Party: Principal Investigator, Tomas Kovarnik, MD, PhD, General University Hospital, Prague
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UK2012; IGA 2012 NT/13224 (Other Grant/Funding Number: Ministry of Health / Czech Republic Grant Agency)
Record Dates: First submitted 2013-01-16; First posted 2013-01-23 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2013-01

CONDITIONS: Coronary Artery Disease
Keywords: Intravascular ultrasound; Virtual histology; Optical coherence tomography; Coronary atherosclerosis; Statins; Retinal imaging
MeSH Terms: conditions — Coronary Artery Disease | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rosuvastatin (Experimental): All patients will be using rosuvastatin 40 mg
  Interventions: Drug: Rosuvastatin

INTERVENTIONS:
Drug: Rosuvastatin — All patients will be using rosuvastatin 40 mg

SUMMARY:
* The prediction of extent and risk profile of coronary atherosclerosis based on clinical evaluation and non-invasive techniques.
* Detailed analysis of plaque volume, plaque composition, risk plaque features and shear stress (WSS) changes during lipid lowering therapy (rosuvastatin 40mg) from 3D vessel reconstruction.
* Prediction of changes in coronary arteries based on changes in non-invasive examinations.
* Examination of WSS influence on atherosclerosis development and changes of WSS during lipid lowering therapy.

DETAILED DESCRIPTION:
The fundamental aim of this project is development of reliable algorithm for detection of extent and risk profile of coronary atherosclerosis based on non-invasive examinations (carotid ultrasound, examination of retinal vessel, diagnosis of endothelial dysfunction, pro-inflammatory markers including new markers of atherosclerosis and gene polymorphisms) with maximal effort on diagnosis of vulnerable plaques. The second part of the study is prediction of coronary atherosclerosis changes during high-dose lipid-lowering therapy (rosuvastatin 40 mg daily). Coronary artery impairment will be examined by up-to date technology using the fusion of angiography, intravascular ultrasound and virtual histology for 3D coronary artery reconstruction together with information about mechanical properties of arteries like a vessel shear stress. This algorithm for non-invasive assessment of coronary impairment and its changes during will be used for detection of high risk patients (in terms of acute coronary syndrome development) and of patients with low response to statin therapy. Further target is detailed assessment of atherosclerosis development and its changes during lipid-lowering therapy.

ELIGIBILITY:
Inclusion Criteria:

* stable angina pectoris

Exclusion Criteria:

* age less than 18 or more than 80
* renal insufficiency
* liver insufficiency
* pregnancy or , child potential without contraception
* intolerance of statins
* rhabdomyolysis or other myopathy in patient´s history
* acute coronary syndrome in last 6 weeks
* coronary anatomy unsuitable for intravascular ultrasound
* active cancer

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-06; Primary Completion 2014-12 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
The prediction of plaque volume and plaque composition. | The patients will be followed in the study for one year
  The study is looking for non-invasive predictors of plaque volume and plaque composition. The non-invasive predictors include carotid ultrasound, polymorphism in gene for heme-oxygenase 1 and retinal imaging.

SECONDARY OUTCOMES:
Prediction of changes in plaque volume and plaque composition | The patients will be followed in the study for one year.
  Prediction of changes in plaque composition and plaque volume during lipid lowering therapy based on changes of non-invasive examination.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (2):
  - Loyola University Hospital, Maywood, Illinois
  - The University of Iowa, Iowa City, Iowa
- General University Hospital, Prague, Czechia

REFERENCES:
- [Background] Kovarnik T, Kral A, Skalicka H, Mintz GS, Kralik L, Chval M, Horak J, Skalicka L, Sonka M, Wahle A, Downe RW, Uhrova J, Benakova H, Cernohousova L, Martasek P, Belohlavek J, Aschermann M, Linhart A. The prediction of coronary artery disease based on non-invasive examinations and heme oxygenase 1 polymorphism versus virtual histology. J Invasive Cardiol. 2013 Jan;25(1):32-7. PMID 23293173
- [Background] Sonka M, Downe RW, Garvin JW, Lopez J, Kovarnik T, Wahle A. IVUS-based assessment of 3D morphology and virtual histology: prediction of atherosclerotic plaque status and changes. Annu Int Conf IEEE Eng Med Biol Soc. 2011;2011:6647-50. doi: 10.1109/IEMBS.2011.6091639. PMID 22255863
- [Derived] Kovarnik T, Chen Z, Mintz GS, Wahle A, Bayerova K, Kral A, Chval M, Kopriva K, Lopez J, Sonka M, Linhart A. Plaque volume and plaque risk profile in diabetic vs. non-diabetic patients undergoing lipid-lowering therapy: a study based on 3D intravascular ultrasound and virtual histology. Cardiovasc Diabetol. 2017 Dec 7;16(1):156. doi: 10.1186/s12933-017-0637-0. PMID 29212544